CLINICAL TRIAL: NCT05295758
Title: ACHIEVE GREATER: Addressing Cardiometabolic Health Inequities by Early PreVEntion in the GREAT LakEs Region
Brief Title: Project 1: ACHIEVE- HTN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due lack of eligible participants
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Robert D Brook, Director, Cardiovascular Prevention Professor of Medicine, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-22-01-4343
Record Dates: First submitted 2022-03-08; First posted 2022-03-25 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Hypertension; Undiagnosed Diseases
Keywords: Health Disparities; African American; Prevention
MeSH Terms: conditions — Hypertension; Undiagnosed Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PAL2 Intervention (Experimental): Overall study cohort will be enrolled into non-randomized active treatment
  Interventions: Behavioral: PAL2

INTERVENTIONS:
Behavioral: PAL2 — Community health worked based intervention to mitigate psychosocial and life circumstance barriers to optimize health promotion coupled with high blood pressure and lifestyle disease state education
  Other Names:
  Pragmatic personalized, adaptable approach to lifestyle and life circumstance

SUMMARY:
This project is part of the ACHIEVE GREATER (Addressing Cardiometabolic Health Inequities by Early PreVEntion in the GREAT LakEs Region) Center (IRB 100221MP2A), the purpose of which is to reduce cardiometabolic health disparities and downstream Black-White lifespan inequality in two cities: Detroit, Michigan, and Cleveland, Ohio. The ACHIEVE GREATER Center will involve three separate but related projects that aim to mitigate health disparities in risk factor control for three chronic conditions, hypertension (HTN, Project 1), heart failure (HF, Project 2) and coronary heart disease (CHD, Project 3), which drive downstream lifespan inequality. All three projects will involve the use of Community Health Workers (CHWs) to deliver an evidence-based practice intervention program called PAL2. All three projects will also utilize the PAL2 Implementation Intervention (PAL2-II), which is a set of structured training and evaluation strategies designed to optimize CHW competence and adherence (i.e., fidelity) to the PAL2 intervention program. The present study is Project 1 of the ACHIEVE GREATER Center

DETAILED DESCRIPTION:
Hypertension (HTN) is the leading risk factor for global morbidity and mortality, accounting for a significant proportion of atherosclerotic cardiovascular disease (CVD), heart failure and chronic kidney disease. Even mild elevations in blood pressure (BP) are harmful whereby individuals with stage 1 HTN (130-139/80-89 mm Hg) are already at double CVD risk. Accordingly, the latest HTN guidelines advocated for earlier treatment to reduce the health consequences and prevent the progression to more severe stages which further increases CVD risk. While nearly half of all Americans have HTN, Black adults suffer from a higher prevalence, worse control rates, and more frequent adverse health effects. They are also at heightened risk for an earlier and accelerated progression from mild to more severe HTN. Unfortunately, little progress has been made over past decades in mitigating health inequities related to high BP. In fact, predominantly Black cities such as Detroit disproportionately suffer from nearly twice the national average mortality rate due to CVD.

Mounting evidence shows that pervasive negative social determinants of heath (SDoH) are major drivers of these inequities and represent a critical barrier to achieving BP control in Black hypertensives. Core issues include poor access to healthcare and a burdensome system for care linkage especially in under-resourced settings, low health education and literacy, and structural inadequacies in care delivery including a failure to address the spectrum of life circumstances that elevate BP and hinder the adoption of salutary lifestyle changes. These systemic issues must be addressed, and remedied early in the hypertension disease process, if the health burden and CVD sequela of high BP are to be successfully reduced in Black communities. To address parallel racial inequities related to COVID-19 in Detroit, we developed an innovative mobile health unit (MHU) program that uses geospatial health and social vulnerability data to target deployment of specially outfitted vehicles to predominately Black communities with the highest needs. Since April 2020, Wayne Health Mobile Unit conducted 550 events with 220 community partners where 45,000 people have been vaccinated or tested for COVID.

In PROJECT 1 (ACHIEVE HTN), of the ACHIEVE GREATER (Addressing Cardiometabolic Health Inequities by Early Prevention in the Great Lakes Region) research center, the project proposes an innovative approach to identify and control HTN at its earliest stages in undiagnosed Black adults, potentially yielding an enormous benefit towards lifetime health equity. Using a hybrid type I effectiveness-implementation and quasi-experimental design, we will leverage our MHU platform to implement a program that links low CVD risk Black adults with stage 1 HTN to collaborative care delivered by non-physicians, community health workers (CHWs) and pharmacists, consisting of a personalized, adaptable approach to lifestyle and life circumstance (PAL2) intervention for 12-months. Core features of PAL2 include the ability to choose from a menu of readily available interventions that address individual negative SDoH, culturally sensitive health and lifestyle education, and adaptability over time according to its acceptance, effectiveness (reduction in home BP), and evolving patient needs. If BP remains ≥130/80 mm Hg after 6 months, a pharmacist-directed medical treatment algorithm will be added to PAL2 to achieve timely BP control. Program benefits, including BP-lowering, will be assessed during implementation (12-months) and maintenance phases (year 2) after linkage to medical care.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, an individual must meet all of the following criteria:

  1. Self-identified Black/African Americans
  2. Detroit-area residents (defined as those who attend attended a Detroit-area community event)
  3. > 18 years of age
  4. Screening systolic BP 130-139 and diastolic BP < 90 mm Hg
  5. Not currently taking medications for HTN (Untreated)
  6. 10-year cardiovascular risk < 10% per ASCVD calculator (as such nearly all patients will be <50-55 years of age)
  7. Baseline home systolic BP 120-159 mm Hg and diastolic BP < 100 mm Hg

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  1. History of clinical cardiovascular disease (CVD)
  2. History of kidney disease or eGFR <60 mL/min from screening labs
  3. Self-reported pregnancy (or planning to be pregnant in the next year)
  4. History of diabetes or HbA1c > 6.5% from SOC screening labs
  5. Non-HDL-C > 220 mg/dL from SOC labs (potential genetic hyperlipidemia)
  6. Arm circumference > 18'' (home BP arm cuff will be inaccurate)
  7. Baseline home BP average > 160mm Hg systolic and/or >100 mm Hg diastolic

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Home systolic blood pressure (BP) | 12 months
  Change in home systolic BP at 12-months versus baseline (detect ≥ 3 mm Hg difference). This will be determined by comparing the "post-trial home systolic BP" (7-day average) versus the "baseline home systolic BP" (7-day average).
Blood pressure control rate | 12 months
  Percentage of study participants who achieve blood pressure control (< 130/80) at 12 months compared to baseline.

SECONDARY OUTCOMES:
BP control without medication use | 12 Months
  1. Effectiveness of the PAL2 intervention will be assessed by the percentage of participants who achieve BP control (<130/80 mm Hg) by lifestyle and PAL2 intervention alone without requiring medication.
Population reach | 12 months
  Reach will be assessed by evaluating the number of patients who are screened by the MHUs; the number and percentage of screened patients who meet inclusion and exclusion criteria for ACHIEVE HTN; the number and percentage of patients who meet inclusion that enroll; and the number and percentage of enrolled patients who do and do not complete the study. For each of these measures, qualitative and quantitative methods will be utilized to understand how patient and community level characteristics may have contributed to higher or lower indicators of reach.
Durability of BP control over 2 years | 24 months
  Durability will be evaluated by the change in systolic BP from 12 months to 24 months.
Home diastolic BP | 12months
  Effect of PAL2 on diastolic BP will be evaluated by the change in diastolic BP from baseline to 12 months.

OTHER OUTCOMES:
Patient wellbeing | 12 months
  Patient satisfaction and impact of the PAL2 intervention on quality of life and wellbeing will be evaluated by questionnaires administered at baseline and month 12.
Cost effectiveness | 12 months
  Cost Effectiveness of the PAL2 intervention will determined using disaggregated cost analysis, assessing the cost of intermediate inputs per endpoint achieved, providing a detailed breakdown of resources used. To allow some cross-intervention benchmarking, we additionally estimate the cost per quality adjusted life years (QALY) extended by the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State, Detroit, Michigan, United States